CLINICAL TRIAL: NCT02742181
Title: A Prospective Randomized Control Trial of The Effectiveness of Entereg as a Rescue Treatment of Postoperative Ileus Following Colorectal Surgery
Brief Title: Alvimopan as Rescue in Post op Ileus
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated due to lack of enrollment
Sponsor: Sharon Stein (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor-Investigator, Sharon Stein, Staff Surgeon, Associate Professor of Surgery, University Hospitals Cleveland Medical Center
Organization: University Hospitals Cleveland Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-15-28
Record Dates: First submitted 2016-04-04; First posted 2016-04-18 (Estimated); Results first posted 2022-11-18 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-10

CONDITIONS: Colorectal Surgery; Ileus
MeSH Terms: conditions — Ileus | interventions — alvimopan; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Alvimopan group (Experimental): In addition to standard postoperative care, patients randomized to the study group will be given 12mg of alvimopan orally twice a day, from the time of diagnosis of postoperative ileus to the time of return of bowel function or for 5 days.
  Interventions: Drug: Alvimopan
- Control Group (Other): Patients randomized to the control group receive standard postoperative care which includes but is not limited to NPO status, IV fluid rehydration, and nasogastric decompression.
  Interventions: Other: Control Group

INTERVENTIONS:
Drug: Alvimopan — Subjects diagnosed with a post operative ileus after surgery will be given alvimopan
  Other Names: Entereg
  Arms: Alvimopan group
Other: Control Group — Standard postoperative care
  Arms: Control Group

SUMMARY:
This will be a prospective randomized control trial with a total of 142 patients. Patients who undergo laparoscopic or open colorectal resection, small bowel resection, or ileostomy reversal with small bowel resection that subsequently develop postoperative ileus will be eligible for enrollment. If they meet inclusion/exclusion criteria, they will be randomized at the time of diagnosis of postoperative ileus to receive Entereg as rescue therapy or to receive conservative standard care.

Patients randomized to the Entereg group will be given 12mg of Entereg two times daily from the time of randomization until the return of bowel function or 5 days. Both groups will be treated with conservative standard care, including bowel rest, reduction in oral diet, and placement of nasogastric tube as clinically indicated.

All patients will follow a standard ERAS pathway after surgery, with early feeding and ambulation, along with opioid minimizing measures as is our standard postoperative protocol.

Primary outcome will be hospital length of stay. Secondary outcomes will include time to return of bowel function, 30-day morbidity/mortality, complications, reoperation and readmission.

Total number of patients: 142 Patients in each study group: 71

DETAILED DESCRIPTION:
At the time of diagnosis of postoperative ileus and after enrollment and randomization, all patients will be returned to NPO status. Nasogastric tubes (NGT) may be placed for gastric decompression at the discretion of the surgical team if clinically indicated. In the event that an NGT is placed, medications will be given orally or via the NGT, which will be clamped for 30 minutes after administration. Patients will continue on standard ERAS pathways with the exception of reduction of diet. Antiemetics will be given as clinically indicated; however, no prokinetic or promotility agents will be given as scheduled dosages.

Patients randomized to the study group will be given 12mg of Entereg orally twice a day, from the time of diagnosis of postoperative ileus to the time of return of bowel function or for 5 days.

Patients randomized to the control group receive standard postoperative care.

The patient and surgical team will be able to know which arm of the study the patient is in based on documentation in the medical record of the administration of Entereg.

Patients in both groups will remain NPO until the return of bowel function, defined as passage of stool, decrease in nasogastric tube output. At this point, the nasogastric tube will be removed and a trial of oral diet will be attempted per surgeon's discretion.

Standard discharge criteria will be applied to all patients, including:

* Passage of stool
* Ability to tolerate solid food and to drink comfortably
* Adequate oral analgesia
* Patient's willingness to be discharged.

Data to be collected The medical/surgical information below will be collected as part of this research study and is all information already available as part of the patients medical chart.

* Patient name, medical record number
* Past Medical History
* Past Surgical history
* Preoperative Medications (including steroids, anticoagulation, opioid use)
* Pre-operative Diagnosis
* Patient Demographics (age, gender, BMI, ASA score)
* Procedure performed
* Time of surgery
* Wound classification
* Estimated blood loss
* Intraoperative transfusion
* Intraoperative IV fluids given
* Conversion from laparoscopic to open procedure
* Stoma creation
* Time/day surgery to ileus
* Time from surgery to medication given
* Time from ileus diagnosis to medication given
* Was there return of bowel function (flatus or stool, solid or liquid, stoma output) prior to ileus
* Intra-abdominal infection/anastomotic leak
* Time/day of return of bowel function post ileus (flatus and stool- solid or liquid, and stoma function)
* Time/day of ability to tolerate oral diet (liquid and solid food)
* Nasogastric tube placement and daily output
* Duration of nasogastric tube
* Use and type of anti-emetics given
* Total number of Entereg doses given
* Post operative complications including reoperation
* Length of stay in hospital, defined as time from surgery to discharge
* 30-day readmissions

Study Completion Completion of participation in the study will be 30 days after the date of surgery. Any readmission up to 30 days post-operatively to the hospital as a direct result of their surgery will be followed. The patients will follow-up with the surgeon in the office in approximately 3-6 weeks, which is considered standard of care for all patients undergoing colorectal surgery and is not considered part of the research study. Any patient for whom follow-up documentation is missing or incomplete shall be contacted via telephone. The purpose of the call will be to simply determine return to function and outcome. Only a co-investigator shall contact the subject and will identify themselves at the beginning of the call. Any subject can reserve the right not to participate in the phone call interview; they would remain in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who have benign or malignant colonic or rectal disease that have undergone laparoscopic or open colorectal resection, small bowel resection or ileostomy reversal with small bowel resection and subsequently developed postoperative ileus, defined as:

   * Return to NPO status after initial diet attempts, or
   * Placement of nasogastric tube
2. Subjects who are 18 years of age and older
3. Subjects of either gender
4. Subjects who are willing and able to adhere to protocol requirements, agree to participate in the study program and provide written and informed consent.

Exclusion Criteria:

1. Subjects who received Entereg preoperatively.
2. Subjects that have taken therapeutic doses of opioids for more than 7 days immediately prior to surgery.
3. Subjects with severe hepatic impairment.
4. Subjects with end-stage renal disease.
5. Subjects who are pregnant.
6. Subjects who were diagnosed with a complete small bowel obstruction preoperatively.
7. Subjects with a medical condition that may interfere with the use of the study medication Entereg.
8. Subjects who have a condition or general disability or infirmity that in the opinion of the investigator precludes further participation in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2015-12-02 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Stein, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Case Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Story SK, Chamberlain RS. A comprehensive review of evidence-based strategies to prevent and treat postoperative ileus. Dig Surg. 2009;26(4):265-75. doi: 10.1159/000227765. Epub 2009 Jul 3. PMID 19590205
- [Background] Bauer AJ, Boeckxstaens GE. Mechanisms of postoperative ileus. Neurogastroenterol Motil. 2004 Oct;16 Suppl 2:54-60. doi: 10.1111/j.1743-3150.2004.00558.x. PMID 15357852
- [Background] Holte K, Kehlet H. Postoperative ileus: a preventable event. Br J Surg. 2000 Nov;87(11):1480-93. doi: 10.1046/j.1365-2168.2000.01595.x. PMID 11091234
- [Background] Behm B, Stollman N. Postoperative ileus: etiologies and interventions. Clin Gastroenterol Hepatol. 2003 Mar;1(2):71-80. doi: 10.1053/cgh.2003.50012. PMID 15017498
- [Background] Luckey A, Livingston E, Tache Y. Mechanisms and treatment of postoperative ileus. Arch Surg. 2003 Feb;138(2):206-14. doi: 10.1001/archsurg.138.2.206. PMID 12578422
- [Background] Delaney CP, Brady K, Woconish D, Parmar SP, Champagne BJ. Towards optimizing perioperative colorectal care: outcomes for 1,000 consecutive laparoscopic colon procedures using enhanced recovery pathways. Am J Surg. 2012 Mar;203(3):353-5; discussion 355-6. doi: 10.1016/j.amjsurg.2011.09.017. Epub 2012 Jan 20. PMID 22264739
- [Background] Zhuang CL, Ye XZ, Zhang XD, Chen BC, Yu Z. Enhanced recovery after surgery programs versus traditional care for colorectal surgery: a meta-analysis of randomized controlled trials. Dis Colon Rectum. 2013 May;56(5):667-78. doi: 10.1097/DCR.0b013e3182812842. PMID 23575408
- [Background] Delaney CP, Wolff BG, Viscusi ER, Senagore AJ, Fort JG, Du W, Techner L, Wallin B. Alvimopan, for postoperative ileus following bowel resection: a pooled analysis of phase III studies. Ann Surg. 2007 Mar;245(3):355-63. doi: 10.1097/01.sla.0000232538.72458.93. PMID 17435541
- [Background] Delaney CP, Craver C, Gibbons MM, Rachfal AW, VandePol CJ, Cook SF, Poston SA, Calloway M, Techner L. Evaluation of clinical outcomes with alvimopan in clinical practice: a national matched-cohort study in patients undergoing bowel resection. Ann Surg. 2012 Apr;255(4):731-8. doi: 10.1097/SLA.0b013e31824a36cc. PMID 22388106
- [Background] Senagore AJ, Bauer JJ, Du W, Techner L. Alvimopan accelerates gastrointestinal recovery after bowel resection regardless of age, gender, race, or concomitant medication use. Surgery. 2007 Oct;142(4):478-86. doi: 10.1016/j.surg.2007.07.004. PMID 17950339
- [Background] Traut U, Brugger L, Kunz R, Pauli-Magnus C, Haug K, Bucher HC, Koller MT. Systemic prokinetic pharmacologic treatment for postoperative adynamic ileus following abdominal surgery in adults. Cochrane Database Syst Rev. 2008 Jan 23;(1):CD004930. doi: 10.1002/14651858.CD004930.pub3. PMID 18254064
- [Background] Zingg U, Miskovic D, Pasternak I, Meyer P, Hamel CT, Metzger U. Effect of bisacodyl on postoperative bowel motility in elective colorectal surgery: a prospective, randomized trial. Int J Colorectal Dis. 2008 Dec;23(12):1175-83. doi: 10.1007/s00384-008-0536-7. Epub 2008 Jul 30. PMID 18665373

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Alvimopan Group | Control Group
Started | 6 | 8
Completed | 5 | 8
Not Completed | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alvimopan Group | Control Group | Total
Number analyzed (Participants) | 6 | 8 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 5 | 7
  >=65 years | 4 | 3 | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 2 | 5 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 4 | 6 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Hospital Length of Stay
Description: Date of surgery until discharge
Time Frame: up to 30 days
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Alvimopan Group | Control Group
Number analyzed (Participants) | 6 | 8
Days | 9 (4.56) | 8.5 (1.48)

2. Secondary Outcome: Time to Return of Bowel Function
Description: Date ileus identified to time of passing flatus, stool and tolerating diet
Time Frame: 30 days
Population: Data not collected
Arm/Group | Alvimopan Group | Control Group
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Complications
Description: All adverse events
Time Frame: 30 days
Measure: Number; unit: Number of AEs
Arm/Group | Alvimopan Group | Control Group
Number analyzed (Participants) | 6 | 8
Number of AEs | 4 | 6

4. Secondary Outcome: Number of Reoperations
Description: Any reoperations within 30 days of surgery
Time Frame: 30 days
Measure: Number; unit: Number of reoperations
Arm/Group | Alvimopan Group | Control Group
Number analyzed (Participants) | 6 | 8
Number of reoperations | 0 | 0

5. Secondary Outcome: Number of Readmissions
Description: Any readmissions within 30 days of surgery
Time Frame: 30 days
Measure: Number; unit: Number of readmissions
Arm/Group | Alvimopan Group | Control Group
Number analyzed (Participants) | 6 | 8
Number of readmissions | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Alvimopan Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/8
Serious Adverse Events (participants affected / at risk) | 1/6 | 1/8
Other Adverse Events (participants affected / at risk) | 3/6 | 5/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvimopan Group (N=6) | Control Group (N=8)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1 (1) — Severe
Recurrent ileu (General disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Alvimopan Group (N=6) | Control Group (N=8)
Bloody NG output (Gastrointestinal disorders) | 0 | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 — Mild
Urinary retention (Renal and urinary disorders) | 0 | 1 (1)
Thrush (General disorders) | 0 | 1 (1)
Hallucinations (Psychiatric disorders) | 0 | 1 (1)
Exacerbation hypertension (General disorders) | 0 | 1 (1)
Acute Kidney injury (Renal and urinary disorders) | 1 (1) | 0
Urinary tract infection (Renal and urinary disorders) | 1 (1) | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-11-17): https://cdn.clinicaltrials.gov/large-docs/81/NCT02742181/Prot_SAP_000.pdf